CLINICAL TRIAL: NCT00550147
Title: An Open-Label Study of Quetiapine Added to Oros Methylphenidate in the Treatment of ADHD and Aggressive Behavior
Brief Title: Quetiapine and Concerta in the Treatment for ADHD and Aggressive Behavior.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0307-31 (IRB#); NCT00198211 (obsolete NCT alias)
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD-Combined TypeDisruptive behavior Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Oros Methylphenidate and Quetiapine
  Interventions: Drug: Oros Methylphenidate; Drug: quetiapine

INTERVENTIONS:
Drug: Oros Methylphenidate — Oros methylphenidate will be titrated over 3 visits according to the following schedule:
  * Visit 2 dose of 18 mg QAM
  * Visit 3 dose of 36mg QAM
  * Visit 4 dose of 54mg QAM.
  Other Names: Concerta
Drug: quetiapine — Quetiapine will be titrated according to the following schedule as determined by efficacy and safety assessments (See Table 1).
  Table 1: Quetiapine Dosing Schedule (subject's required weight = 30-80 kg)
  * Visit 5 dose of 25mg BID
  * Visit 6 dose of 50mg BID
  * Visit 7 dose of 100mg BID
  * Visit 8 dose of 200mg BID
  * Visit 9 dose of 300mg BID
  Efficacy: For any visit following Visit 5, dosage will remain stable if clinically significant improvement criteria are met.If subjects subsequently fail to meet clinically significant improvement criteria, dose increases will resume at the next level of the dosing schedule.
  Other Names: Seroquel

SUMMARY:
The primary purpose of this thirteen-week, open-label study is to test the hypothesis that quetiapine in combination with Oros methylphenidate will reduce aggressive symptoms in children and adolescents who have shown inadequate response to OROS methylphenidate alone.

DETAILED DESCRIPTION:
Informed consent will be obtained from the subject and parent or legal guardian before any study procedures begin. Study procedures will include the verification of inclusion and exclusion criteria, and completion of assessments and safety measures (physical examination, vital signs, adverse events and concomitant medication review, AIMS, laboratory tests, ECG, pregnancy test) as indicated in the Schedule of Events. All laboratory and electrocardiogram results must be reviewed by a physician before the subject returns for Visit 2.

Study Period II (Visits 2-5)

All subjects meeting entry criteria will initially receive Oros methylphenidate beginning at Visit 2. The Oros methylphenidate will be titrated over 3 visits according to the following schedule:

* Visit 2 dose of 18 mg QAM
* Visit 3 dose of 36mg QAM
* Visit 4 dose of 54mg QAM.
* At Visit 5, any subjects unable to tolerate continuation of the Oros methylphenidate dose of 54mg QAM or subjects that meet improvement criteria as defined above will be discontinued from the study. Subjects able to tolerate the daily dose of 54mg Oros methylphenidate and who do not meet improvement criteria at Visit 5 will begin receiving quetiapine in addition to continuing Oros methylphenidate at 54mg QAM for the balance of the study. The initial dose of quetiapine dispensed at Visit 5 will be 25mg QAM for one day with an increase to 25mg BID until Visit 6.

At each visit safety and efficacy information will be completed according to the Schedule of Events.

Study Period III (Visits 6-10) Quetiapine will be titrated at Visits 6 - 9 according to the parameters in the quetiapine dosing schedule and the completion of safety and efficacy measures listed in the Schedule of Events. A telephone follow-up with the parent or legal guardian will be made 7-9 days after Visit 8 for physician review of subject adverse events and safety.

At visit 10 subjects will be given clinical recommendations for follow-up care from a physician investigator after completion of all study procedures (labs/EKG, vital signs, physical exam, AIMS, ADHD-RS-IV, CGI-I, CGI-S, RAAPP, MOAS, SNAP, CCPT)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 12 yrs.old but less than 18 when informed consent is obtained.
2. Subjects must meet DSM-IV criteria for ADHD/Combined Type and one of the Disruptive Behavior Disorders as diagnosed by clinical interview and confirmed by the Kiddie-SADS-PL (K-SADS-PL) semistructured diagnostic interview.
3. Subjects must have one DSM-IV aggressive feature of Conduct Disorder (CD) as rated on the K-SADS-PL including:

   * initiation of physical fights (CD symptom A2)
   * use of a weapon to bring harm to others (CD symptom A3)
   * physical cruelty to people (CD symptom A4) or animals (CD symptom A5)
   * confrontation stealing (CD symptom A6)
   * destruction of property (CD symptom A8 or A9).
4. Subjects must have severe aggressive and ADHD symptoms as indicated by a global CGI score of 4 or greater and a RAAPP score of 4 or 5 at Visit 1.
5. Subjects must have had at least four outbursts per month involving destruction of property, verbal aggression, or physical aggression toward others or self during the past two months at Visit 1.
6. Subjects with previous trials of psychostimulants must have had a response insufficient to markedly change overall quality of life as defined by a CGI score of 3 or greater based on interview with the parent.
7. Subjects must not have taken any medication for the treatment of ADHD or DBD for either 5 half-lives of the medication or 28 days (whichever is less) at Visit 1. If subjects are currently taking medications for the treatment of ADHD or DBD, the assent and consent must be reviewed and signed by the subject and parent/legal guardians (Visit 0) before the physician investigator will provide a tapering schedule for current medications.
8. Laboratory results obtained at Visit 1 must be reviewed by a physician by Visit 2 and show no significant abnormalities.
9. Baseline electrocardiogram (ECG) results obtained at Visit 1 must be assessed by a physician by Visit 2 and show no significant abnormalities.

Exclusion Criteria:

1. Subjects with likely mental retardation as defined as a K-BIT Matrices IQ score of less than 70 at Visit 1.
2. Subjects who meet criteria for bipolar disorder as diagnosed by clinical interview and confirmed by the K-SADS-PL at Visit 1.
3. Subjects with a biological parent or sibling who meets criteria for bipolar disorder.
4. Subjects who have any history of psychosis.
5. Subjects who weigh less than 30kg or more than 80kg at study entry.
6. Female subjects who are pregnant or who are breast-feeding as assessed at Visit 1.

   Postmenarcheal sexually-active females who are not using a clinically acceptable method of birth control.
7. Subjects with a history of any seizure disorder other than febrile seizures.
8. Subjects with a history of alcohol or drug abuse within the past three months or who are currently using alcohol, drugs of abuse, or any prescribed or over-the-counter medications in a manner considered abusive by the investigators.
9. Subjects currently taking any psychotropic medications or who are likely to need psychotropic medications during the study as assessed by the physician at Visit 1.
10. Subjects considered to be at serious suicidal risk.
11. Subjects taking any medications that are not reviewed and approved by a physician investigator. Specific requirements include:

    * Psychotropic medications other than quetiapine and Concerta may not be used during the trial.
    * Patients may receive lorazepam or chlorpromazine if needed for severe aggression. These drugs should not be given beyond 24 hours.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2004-02; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Dunn, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Childrens Hospital, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited during the time period 2004-2005, using flyers and letters sent to local schools, clinics, and community agencies, as well as from referrals to the site at which the study was conducted.
Pre-assignment Details: All eligible subjects were assigned to the first phase of treatment (Oros MPH alone).
Groups:
- OROS Methylphenidate and Quetiapine: This is the Baseline Visit, immediately after enrollment and prior to taking any medication. All enrolled subjects start taking OROS methylphenidate until Visit 5. At visit 5, if there is significant improvement (decrease in aggressive symptoms), then subject is discontinued from the study. If there is not significant improvement, then subject continues in study and begins taking OROS methylphenidate plus quetiapine. 24 of 30 subjects entered the OROS methylphenidate and quetiapine arm. 4 subjects made significant improvement at visit 5 and were discontinued from the study; 2 subjects were withdrawn from the study prior to visit 5. Therefore, 6 of 30 subjects did not enter the OROS methylphenidate and quetiapine arm. Only 24 of 30 subjects entered this arm. Visit 10 is measured at the end of OROS MPH+Quetiapine treatment
Period: OROS Methylphenidate Monotherapy
Arm/Group | OROS Methylphenidate and Quetiapine
Started | 30
Completed | 24
Not Completed | 6
Not completed — significant improvement at visit 5 | 4
Not completed — Withdrawal by Subject | 2
Period: Quetiapine Addition Treatment Period
Arm/Group | OROS Methylphenidate and Quetiapine
Started | 24
Completed | 18
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Noncompliance | 2
Not completed — Moved out of state | 1

BASELINE CHARACTERISTICS:
Groups:
- OROS Methylphenidate and Quetiapine: All enrolled subjects start taking OROS methylphenidate. At visit 5, if there is significant improvement (decrease in aggressive symptoms), then subject is discontinued from the study. If there is not significant improvement, then subject continues in study and begins taking OROS methylphenidate plus quetiapine. Therefore enters the OROS methylphenidate and quetiapine arm. 24 of 30 subjects entered the OROS methylphenidate and quetiapine arm. 4 subjects made significant improvement at visit 5 and were discontinued from the study, and, therefore, did not enter the OROS methylphenidate and quetiapine arm. 2 subjects were withdrawn from the study prior to visit 5, and, therefore, did not enter the OROS methylphenidate and quetiapine arm. Therefore, 6 of 30 subjects did not enter the OROS methylphenidate and quetiapine arm. Only 24 of 30 subjects entered this arm.
Arm/Group | OROS Methylphenidate and Quetiapine
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.2 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: RAAPP: Rating of Aggression Against People and/or Property Scale
Description: The RAAPP is a global rating scale of aggression that is completed by a clinician based on interview and observation data. It is scored from 1 (no aggression reported) to 5 (intolerable behavior).
Time Frame: See Arm/Group - Repeated Measures
Population: Participants were those who qualified for the augmentation portion of the study (inadequate response to Oros MPH alone). Analysis was per protocol (intent-to-treat, LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline: Baseline score at study entry
- Visit 5 - MPH Monotherapy - Week 4: Score following treatment with MPH monotherapy after Week 4
- Visit 10 - MPH+Quetiapine - Week 13: Score following treatment with combined MPH and quetiapine after Week 13
Arm/Group | Baseline | Visit 5 - MPH Monotherapy - Week 4 | Visit 10 - MPH+Quetiapine - Week 13
Number analyzed (Participants) | 24 | 24 | 24
units on a scale | 4.3 (0.4) | 3.2 (0.6) | 2.0 (0.8)
Statistical Analysis 1: Comparison: Visit 5 - MPH Monotherapy - Week 4 vs Visit 10 - MPH+Quetiapine - Week 13; This was a repeated-measures analysis, using a single group of subjects who were administered quetiapine in addition to OROS mph. See Kronenberger et al. (2007, Journal of Child and Adolescent Psychopharmacology) for additional information; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Paired t-test (comparing augmentation period start score with end score), 23 df. Value is Visit 10 score minus Visit 5 score (null hypothesis=0); Mean Difference (Final Values) = -1.125, 95% CI 2-sided [-1.52 to -0.72], Standard Error of Mean 0.1933 — This was a comparison of pre-post change in a single group, with treatment administered open-label

2. Secondary Outcome: CGI-S: Clinical Global Improvement Scale
Description: The CGI-S is a 1-7 investigator rating of overall severity of target behavioral symptoms, which will be completed at each visit as a secondary efficacy measure of global behavioral functioning. A score of 1 indicates "normal, not ill at all" and a score of 7 indicates "among the most extremely ill patients".
Time Frame: See Arm/Group - Repeated Measures
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline: Baseline scores at study entry
- Visit 10 - MPH + Quetiapine - Week 13: Score following treatment with MPH+quetiapine after Week 13
Arm/Group | Baseline | Visit 5 - MPH Monotherapy - Week 4 | Visit 10 - MPH + Quetiapine - Week 13
Number analyzed (Participants) | 24 | 24 | 24
units on a scale | 5.3 (0.6) | 4.1 (0.8) | 2.8 (0.9)
Statistical Analysis 1: Comparison: Visit 5 - MPH Monotherapy - Week 4 vs Visit 10 - MPH + Quetiapine - Week 13; This was a repeated-measures analysis, using a single group of subjects who were administered quetiapine in addition to OROS mph. Results reported here are for the augmentation period (Visit 5-10). See Kronenberger et al. (2007, Journal of Child and Adolescent Psychopharmacology) for additional information; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.33, 95% CI [-1.75 to -0.91], Standard Error of Mean 0.2056 — This was a comparison of pre-post change in a single group, with treatment administered open-label

3. Secondary Outcome: Modified Overt Aggression Scale (MOAS)
Description: The Modified Overt Aggression Scale (MOAS) is a clinician-rated scale of aggressive outbursts experienced in the past week. Weightings are assigned for severity and frequency of aggression. MOAS total severity score will be completed as a secondary efficacy measure of aggressive behavior. The range for the MOAS is 0-235. A score of 0 indicates "no aggression" and a score of 235 indicates "the most severe and frequent aggressive outbursts".
Time Frame: See arm/group - repeated measures
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | Visit 5 - MPH Monotherapy - Week 4 | Visit 10 - MPH + Quetiapine - Week 13
Number analyzed (Participants) | 24 | 24 | 24
units on a scale | 229.0 (194.3) | 73.7 (57.9) | 26.3 (33.0)
Statistical Analysis 1: Comparison: Visit 5 - MPH Monotherapy - Week 4 vs Visit 10 - MPH + Quetiapine - Week 13; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -47.3, 95% CI [-74.3 to -20.2], Standard Error of Mean 13.06 — This was a comparison of pre-post change in a single group, with treatment administered open-label

4. Secondary Outcome: Swanson, Nolan and Pelham IV (SNAP-IV) Oppositional-Defiant Disorder Subscale
Description: The Swanson, Nolan and Pelham (SNAP-IV) is a 90-item, parent-completed questionnaire consisting of symptoms of ADHD, aggression, depression, and mania. Parents rate each item from 0(not at all) to 3 (very much) based on their child's behavior during the past week. The scores from the Oppositional-Defiant Disorder section of this questionnaire will be used as secondary efficacy measures of parent-reported aggressive behavior. These scores range from 0-24.
Time Frame: See arm/group - repeated measures analysis
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Visit 10 - MPH+Quetiapine - Week 13: Score following treatment with MPH+quetiapine after Week 13
Arm/Group | Baseline | Visit 5 - MPH Monotherapy - Week 4 | Visit 10 - MPH+Quetiapine - Week 13
Number analyzed (Participants) | 24 | 24 | 24
units on a scale | 19.0 (4.1) | 14.5 (6.2) | 10.3 (6.5)
Statistical Analysis 1: Comparison: Visit 5 - MPH Monotherapy - Week 4 vs Visit 10 - MPH+Quetiapine - Week 13; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.17, 95% CI 2-sided [-7.04 to -1.29], Standard Error of Mean 1.39 — This was a comparison of pre-post change in a single group, with treatment administered open-label

5. Secondary Outcome: Attention Deficit/Hyperactivity Disorder Rating Scale -IV- Parent Version (ADHDRS-IV-Parent Version)
Description: The Attention Deficit/Hyperactivity Disorder Rating Scale -IV- Parent Version (ADHDRS-IV-Parent:Inv) (Faries, Yalcin, Harder, & Heiligenstein, 2001) is an interviewer-administered semi structured interview with the parent, focusing on the 18 DSM-IV symptoms. Ratings are made on a 0 (never or rarely) to 3 (very often) scale. The range of the ADHDRS-IV is 0-54. A zero (0) scores indicates no ADHD symptoms and 54 indicates most severe ADHD symptoms. The ADHDRS-IV-Parent:Inv provides an overall severity score, symptom count, and ADHD diagnosis for the child.
Time Frame: See Arm/Group - repeated measures
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | Visit 5 - MPH Monotherapy - Week 4 | Visit 10 - MPH+Quetiapine - Week 13
Number analyzed (Participants) | 24 | 24 | 24
units on a scale | 45.7 (5.8) | 32.7 (10.8) | 19.4 (9.6)
Statistical Analysis 1: Comparison: Visit 5 - MPH Monotherapy - Week 4 vs Visit 10 - MPH+Quetiapine - Week 13; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.29, 95% CI [-17.76 to -8.82], Standard Error of Mean 2.16 — This was a comparison of pre-post change in a single group, with treatment administered open-label

ADVERSE EVENTS:
Arm/Group | OROS Methylphenidate and Quetiapine
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 23/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OROS Methylphenidate and Quetiapine (N=24)
repiratory illness (Respiratory, thoracic and mediastinal disorders) | 9 (9)
headache (General disorders) | 4 (4)
fatigue/sedation (General disorders) | 12 (12)
reduced appetite (Metabolism and nutrition disorders) | 4 (4)
difficulty sleeping (General disorders) | 7 (7)
stomachache/nausea (Gastrointestinal disorders) | 7 (7)
vomiting (Gastrointestinal disorders) | 4 (4)
flu-like syndrome (General disorders) | 5 (5)
lability/irritability (General disorders) | 4 (4)
bruises/cuts/bumps (Skin and subcutaneous tissue disorders) | 3 (3)
dizziness (General disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
There were no unanticipated limitations/caveats. All of the typical caveats of open-label studies apply: As a result, bias, placebo effects, demand characteristics, and other non-treatment related effects may have contributed to results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No